CLINICAL TRIAL: NCT02424123
Title: Is Protein S100B a Predictor of First-to-chronic Seizure Conversion in Adults? A Prognostic Cohort Study
Brief Title: Is Protein S100B a Predictor of First-to-chronic Seizure Conversion in Adults?
Acronym: SeizS100B
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2014/ET-02; 2015-A00157-42 (Other: RCB number)
Record Dates: First submitted 2015-04-20; First posted 2015-04-22 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Epilepsy; Seizures, Epileptic
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Processing of blood samples: 4-5ml of the blood sample will be centrifuged to isolate serum; S100B, IL-1b, IL-6, NSE levels will be investigated at D0 (T0+6h, T0+12h where T0 is seizure time) D14-D28. The remaining blood and cells will be stored at -80°C for future analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: The study population is composed of patients between 18 and 60 years of age, of both sexes, recruited during consultations for a first epileptic seizure at the emergency department of Nîmes and Marseille Hospitals (CHRU).

SUMMARY:
Seizures represent an important clinical problem, accounting for at least 40% of adult onset epilepsy. Predicting seizure recurrence in subjects experiencing a first seizure is difficult due to the lack of prognostic biomarkers. Recent evidence has indicated that blood-brain barrier (BBB) dysfunction constitutes an etiological factor to seizures. In particular, it has been shown that modification of BBB permeability is associated with seizure activity. In addition, it was demonstrated that BBB permeability can be assessed by measuring serum level of the protein S100B. Based on these data and considerations the investigators will test whether the extent of BBB damage at time of first seizure is predictive for seizure recurrence.

The main objective of this study is to evaluate the association between the absolute (ng/ml) serum S100B levels (measured at time of the first seizure) and the experience, or not, of seizure recurrence within one year of follow-up.

DETAILED DESCRIPTION:
The secondary objectives of this study are to investigate the:

A) Prognostic capacity of serum S100B levels to predict seizure recurrence. B) Association between the variation (%) of serum S100B levels between first seizure episode and scheduled follow-up (D14-D28) and seizure recurrence.

C) Correlation of S100B with IL-1b, IL-6, NSE serum levels at the same time points.

D) Association of serology data with: a) EEG profile (normal/abnormal); b) recurrence of seizures (Y/N).

E) Comparison of S100B serum levels in lesional vs non-lesional patients. F) Establishment of a bio-bank (serum and cells).

ELIGIBILITY:
Inclusion Criteria:

* The patient has been correctly informed.
* The patient must have given his informed and signed consent.
* The patient must be insured or beneficiary of a health insurance plan.
* The patient is at least (≥) 18 years old and less than (<) 60 years old.
* The patient has experienced a first generalized, epileptic seizure (patients with partial onset and secondary generalization can also be included).
* The seizure has occurred less than 24 hours ago.

Exclusion Criteria:

* The patient is participating in another study that may interfere with the results or conclusions of this study.
* Within the past three months, the patient has participated in another study that may interfere with the results or conclusions of this study.
* The patient is in an exclusion period determined by a previous study.
* The patient is under judicial protection.
* The patient refuses to sign the consent.
* It is impossible to correctly inform the patient.
* The patient is pregnant or breast-feeding (MRI contraindicated).
* Patient has a previous abnormal brain imaging (MRI).
* Patient has abnormal biological tests for toxicology (alcohol, cocaine and cannabis tests), blood ionogram (hyponatremia <130mM), liver enzymes (>5N), inflammatory syndrome (elevated C-reactive protein).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population is composed of patients between 18 and 60 years of age, of both sexes, recruited during consultations for a first epileptic seizure at the emergency department of Nîmes and Marseille Hospitals (CHRU).
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Serum S100B level | Day 0 (T0+6 hours)
  ng/ml
Serum S100B level | Day 0 (T0+12 hours)
  ng/ml
Seizure recurrence within 1 year | 12 months
  yes/no

SECONDARY OUTCOMES:
Serum S100B level | Between days 14 and 28
  ng/ml
Serum S100B level | 6 months
  ng/ml
Serum S100B level | 12 months
  ng/ml
Serum S100B level | at time of 2nd seizure (expected max of 12 months)
  ng/ml
Serum IL-1b level | Day 0 (T0+6 hours)
  pg/mL
Serum IL-1b level | Day 0 (T0+12 hours)
  pg/mL
Serum IL-1b level | Between days 14 and 28
  pg/mL
Serum IL-6 level | Day 0 (T0+6 hours)
  pg/mL
Serum IL-6 level | Day 0 (T0+12 hours)
  pg/mL
Serum IL-6 level | Between days 14 and 28
  pg/mL
Serum NSE level | Day 0 (T0+6 hours)
  µg/dL
Serum NSE level | Day 0 (T0+12 hours)
  µg/dL
Serum NSE level | Between days 14 and 28
  µg/dL
Electro encephalogram profile | Day 0
Electro encephalogram profile | Between days 14 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Marchi, MD, Study Director — Institut de Génomique Fonctionnelle, CNRS, Montpellier
Locations (2):
- France (2):
  - APHM - Hôpital Nord, Marseille
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes